CLINICAL TRIAL: NCT02668185
Title: Neurokinin 3 Receptor Antagonism as a Novel Treatment for Menopausal Hot Flushes
Brief Title: Neuropeptide Treatment for Hot Flushes During the Menopause
Acronym: NK3R
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); AstraZeneca (Industry); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15HH2867
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Menopausal Flushing
Keywords: Menopausal flushing
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active drug first (Experimental): Baseline period - 2 weeks NK3R antagonist - AZD4901 - 40mg bd - 4 weeks Washout period - 2 weeks Matched placebo orally bd - 2 weeks Monitoring period - 2 weeks
  Interventions: Drug: NK3R antagonist - AZD4901
- Placebo (Placebo Comparator): Baseline period - 2 weeks Matched placebo orally bd - 2 weeks Washout period - 2 weeks NK3R antagonist - AZD4901 - 40mg bd - 4 weeks Monitoring period - 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NK3R antagonist - AZD4901 — Neurokinin 3 receptor antagonist
  Other Names: nil others
  Arms: Active drug first
Drug: Placebo — Placebo
  Other Names: nil others
  Arms: Placebo

SUMMARY:
Placebo-controlled, double-blinded, cross-over clinical trial of a new investigational product

DETAILED DESCRIPTION:
Double-blinded, placebo-controlled, 2-way crossover study in 30 menopausal women with untreated hot flushes treated with a neurokinin 3 receptor (NK3R) antagonist

Aims:

To investigate whether an NK3R antagonist can reduce menopausal flushing

Treatment:

4 weeks administration of active drug and placebo in random order

ELIGIBILITY:
Inclusion Criteria:

* Menopausal women (≥12 months since last menstrual period or bilateral oophorectomy or with a follicle stimulating hormone (FSH) level ≥20 milli-international units/millilitre (mIU/mL) and an estradiol level <190pmol/l in the absence of a reliable menstrual marker (hysterectomy with ovarian preservation or endometrial ablation)) aged 40-62 years with >7 hot flushes/day some of which are reported as severe or bothersome who have not been on treatment for menopausal symptoms for the preceding 8 weeks.

Exclusion Criteria:

1. Significant illness, as judged by the Investigator, within 2 weeks of first study visit.
2. Volunteer has clinical, laboratory, or electrocardiogram (ECG) evidence of uncontrolled hypertension (defined as systolic blood pressure of ≥ 160 mmHg and/or diastolic blood pressure of ≥100 mmHg); uncontrolled diabetes; or significant pulmonary, renal, hepatic, endocrine, or other systemic disease in the opinion of the Investigator.
3. Participant has a history of Gilbert's syndrome, infectious hepatitis, or other significant hepatic disease (e.g. chronic hepatitis, cirrhosis, autoimmune hepatitis, primary sclerosing cholangitis, non-alcoholic steatohepatitis, or hereditary liver disease) in the opinion of the Investigator.
4. Participant has a history of surgery which in the opinion of the investigator could cause malabsorption (e.g. gastric or small intestinal surgery or gastric bypass surgery or banding), or patient has a disease that causes malabsorption.
5. Clinically significant abnormal ECG and/or abnormalities in ECG at screening as judged by the Investigator.
6. A marked prolongation of QT/corrected QT (QTc) interval (e.g. repeated demonstration of a QTc interval > 450 ms).
7. Confirmed history of ischaemic heart disease.
8. Past (within 1 year of enrollment) or present alcohol or substance abuse
9. Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within at least 3 months of the first administration of AZD4901 in this study. The period of exclusion begins 3 months after the final dose. (Note: patients consented and screened, but not randomised in a previous study are not excluded.)
10. Participant has a history of neoplastic disease within 5 years prior to signing informed consent or is currently on ongoing treatment to prevent cancer recurrence.
11. Involvement in the planning and/or conduct of the study (applies to any AstraZeneca employee and their close relatives and/or staff at the study site directly involved in the study, regardless of their role in accordance with their internal procedures)
12. Inability to understand or cooperate with the requirements of the study
13. Participant is legally or mentally incapacitated
14. Participant has significant psychiatric disease or treatment for psychiatric disease e.g. selective serotonin re-uptake inhibitors (SSRIs) which in the opinion of the Investigator may influence the results of the study.
15. Participant has abnormal screening laboratory values as per the guidelines listed below or other clinically significant, unexplained laboratory abnormality according to the Investigator:

    * Aspartate aminotransferase (AST) >1.5 times upper limit of normal (ULN)
    * Alanine aminotransferase (ALT) > 1.5 times ULN
    * Total bilirubin >1.5 times ULN
    * Serum creatinine >2.0 times ULN
16. Clinically relevant disease and abnormalities (past or present), which in the opinion of the Investigator, may either put the patient at risk to participate in this study or may influence the results of the study or the patient's ability to participate in the study.
17. Participant has a history of hyperthyroidism or hypothyroidism or abnormal screening thyroid tests, as judged by the Investigator. Patients with hypothyroidism who are stable on treatment with normal thyroid function tests may be included in the study if in the opinion of the Investigator this will not influence the results of the study.
18. Participant has seizures, patients with history of seizures or with conditions that increase the risk of seizures.
19. Participant has a history of hypersensitivity to more than 2 chemical classes of drugs, including prescription and over-the-counter medications.
20. Participant has taken any potent or moderate CYP3A4 or CYP2C9 inhibitors, potent or moderate CYP3A4 or CYP2C9 inducers, hormonal contraceptives, antiandrogenic drugs, or other medications specified for the time frame

Ages: 40 Years to 62 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Menopausal women (≥12 months since last menstrual period or bilateral oophorectomy or with a follicle stimulating hormone (FSH) level ≥20 milli-international units/millilitre (mIU/mL) and an estradiol level <190pmol/l in the absence of a reliable menstrual marker (hysterectomy with ovarian preservation or endometrial ablation)) aged 40-62 years with >7 hot flushes/day some of which are reported as severe or bothersome who have not been on treatment for menopausal symptoms for the preceding 8 weeks.
Enrollment: 37 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Waljit S Dhillo, MBBS PhD, Principal Investigator — Imperial College and NHS Trust
Locations (1):
- NIHR/Wellcome Trust Imperial CRF, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prague JK, Abbara A, Comninos AN, Jayasena CN, Higham CE, Adaway J, Keevil BG, Veldhuis JD, Dhillo WS. Neurokinin 3 Receptor Antagonists Do Not Increase FSH or Estradiol Secretion in Menopausal Women. J Endocr Soc. 2019 Nov 14;4(2):bvz009. doi: 10.1210/jendso/bvz009. eCollection 2020 Feb 1. PMID 32318647
- [Derived] Prague JK, Roberts RE, Comninos AN, Clarke S, Jayasena CN, Mohideen P, Lin VH, Stern TP, Panay N, Hunter MS, Webber LC, Dhillo WS. Neurokinin 3 receptor antagonism rapidly improves vasomotor symptoms with sustained duration of action. Menopause. 2018 Aug;25(8):862-869. doi: 10.1097/GME.0000000000001090. PMID 29533369
- [Derived] Prague JK, Roberts RE, Comninos AN, Clarke S, Jayasena CN, Nash Z, Doyle C, Papadopoulou DA, Bloom SR, Mohideen P, Panay N, Hunter MS, Veldhuis JD, Webber LC, Huson L, Dhillo WS. Neurokinin 3 receptor antagonism as a novel treatment for menopausal hot flushes: a phase 2, randomised, double-blind, placebo-controlled trial. Lancet. 2017 May 6;389(10081):1809-1820. doi: 10.1016/S0140-6736(17)30823-1. Epub 2017 Apr 3. PMID 28385352

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Drug First Then Placebo: 2 week baseline period First NK3R antagonist - AZD4901 - 40mg orally bd - for 4 weeks intervention then 2 weeks washout period then second intervention with Matched placebo orally bd for 4 weeks with 2 weeks monitoring period
- Placebo First Then Active Drug: 2 week baseline period First intervention is Placebo - 40mg bd - for 4 weeks, then 2 weeks washout period, then second intervention with NK3R antagonist - AZD4901 - 40mg orally bd - for 4 weeks with 2 weeks monitoring period
Period: Baseline Period (2 Weeks)
Arm/Group | Active Drug First Then Placebo | Placebo First Then Active Drug
Started | 20 | 17
Completed | 20 | 17
Not Completed | 0 | 0
Period: First Intervention (4 Weeks)
Arm/Group | Active Drug First Then Placebo | Placebo First Then Active Drug
Started | 20 | 17
Completed | 18 | 17
Not Completed | 2 | 0
Not completed — Physician Decision | 2 | 0
Period: Washout Period (2 Weeks)
Arm/Group | Active Drug First Then Placebo | Placebo First Then Active Drug
Started | 18 | 17
Completed | 17 | 15
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 2
Period: Second Intervention (4 Weeks)
Arm/Group | Active Drug First Then Placebo | Placebo First Then Active Drug
Started | 17 | 15
Completed | 16 | 12
Not Completed | 1 | 3
Not completed — Physician Decision | 1 | 3
Period: Moitoring Period (2 Weeks)
Arm/Group | Active Drug First Then Placebo | Placebo First Then Active Drug
Started | 16 | 12
Completed | 16 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: Crossover study - all participants
Arm/Group | Overall Participants
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 17
  White European | 2
  White Other | 1
  White Unspecified | 1
  Asian, Pakistani | 1
  Black Carribean | 5
  Mixed white and black carribean | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 37

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Hot Flushes During the Final Week of Each 4 Weeks Treatment Period
Description: To ensure accurate records, participants recorded their flushes in real time using either a tally chart on a piece of paper (n=34) or an application on their smartphone such as Tally Counter (Pixel Research Labs, Minneapolis-Saint Paul, MN, USA; n=3), and then collated their total number of flushes twice daily on waking to record previous overnight symptoms and before bed to record daytime symptoms.
Time Frame: Final week of each 4 week treatment period
Population: Whole group intention to treat analysis irrespective of treatment assignment order, adjusted means from crossover analysis with 95% CIs: percentage change in total no. hot flush frequency during final week of 4 week treatment period with MLE4901 and placebo vs with total no. hot flush frequency during the final week of the 2 week baseline period.
Measure: Mean (95% Confidence Interval); unit: hot flushes
Groups:
- Active Drug: NK3R antagonist - AZD4901 - 40mg bd - for 4 weeks
  NK3R antagonist - AZD4901: Neurokinin 3 receptor antagonist
- Placebo: Placebo - 40mg bd - for 4 weeks
  Placebo: Placebo
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 28 | 28
hot flushes | 19.35 [15.99 to 23.42] | 49.01 [40.81 to 58.56]
Statistical Analysis 1: Comparison: Active Drug vs Placebo; Test type: Superiority — Generalised linear mixed model with a Poisson error structure; p < 0.0001, generalised linear mixed model with a Po — Intention to treat adjusted means; Adjusted for intention to treat; Mean Difference (Net) = 29.66, 95% CI 2-sided [17.39 to 42.87]

2. Secondary Outcome: Hot Flush Severity
Description: Score on a scale - HF severity (rated as 1-nil, 2-mild, 3-moderate, 4-severe, as per Joffe 2014) recorded twice daily (day/night as described above for HF frequency). Scores are summed.
Time Frame: Twice daily, morning and night for 14 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: numerical rating of severity by particip
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 28 | 28
numerical rating of severity by particip | 3.27 [2.92 to 3.66] | 5.70 [5.09 to 6.38]
Statistical Analysis 1: Comparison: Active Drug vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = 50

3. Secondary Outcome: Hot Flush Bother
Description: Score on a scale - HF bother (rated as 1-none, 2-a little, 3-moderate, 4-a lot, as per Joffe 2014) will be recorded twice daily (day/night as described above for HF frequency). The data will be analysed as detailed above for the HF frequency. Scores are summed.
Time Frame: twice daily (day/night) for 14 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 28 | 28
score on a scale | 2.92 [2.61 to 3.27] | 5.56 [4.96 to 6.27]
Statistical Analysis 1: Comparison: Active Drug vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis

4. Secondary Outcome: Hot Flush Interference
Description: Score on a scale Menopause Specific Quality of Life (MENQOL) questionnaire 0=not bothered at all - 6=extremely bothered. 4 domains, mean calculated for set of questions in each domain. Overall score is a mean of the means. Highr scor = higher interference.
Time Frame: Daily at bedtime for 14 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Score by participant on 'interference sc
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 28 | 28
Score by participant on 'interference sc | 7.94 [5.76 to 10.95] | 26.48 [20.02 to 35.03]
Statistical Analysis 1: Comparison: Active Drug vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis

5. Secondary Outcome: Skin Conductance Monitor Data.
Description: Mean number of flushes detected during the 48 hours by the skin conductance monitoring will be compared each week when the patients receive AZD4901 versus placebo
Time Frame: Once per week for 48 hours over 14 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of hot flushes detected by monito
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 28 | 28
Number of hot flushes detected by monito | 16.22 [13.99 to 18.8] | 26.91 [23.16 to 31.27]
Statistical Analysis 1: Comparison: Active Drug vs Placebo; Test type: Superiority; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Active Drug First Then Placebo | Placebo First Then Active Drug
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 3/28 | 0/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Drug First Then Placebo (N=28) | Placebo First Then Active Drug (N=28)
transaminase elevations by treatment and CTCAE grade (Hepatobiliary disorders) | 3 (3) | 0 (0) — transient transaminase rise (alanine aminotransferase [ALT] greater than aspartate aminotransferase [AST]) with a normal bilirubin following treatment with MLE4901

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes